CLINICAL TRIAL: NCT00400517
Title: Phase II Trial of Neoadjuvant GM-CSF + Thalidomide in High-Risk Patients With Prostate Cancer Undergoing Prostatectomy
Brief Title: GM-CSF and Thalidomide in Treating Patients Undergoing Surgery for High-Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-4643; P30CA043703 (NIH); CASE-CCF-4643 (Other: Case Comprehensive Cancer Center); CELGENE-CASE-CCF-4643 (Other: Sponsor); BRLX-CASE-CCF-4643 (Other: Sponsor)
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; stage II prostate cancer; adenocarcinoma of the prostate; stage I prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Thalidomide; Neoadjuvant Therapy

ARMS (1):
- GM-CSF Injections and Oral Thalidomide (Experimental): taught to administer an injection of GM-CSF under your skin (subcutaneous injection) and will administer this medicine to yourself every Monday, Wednesday and Friday for 4 weeks at time. Thalidomide will be taken orally (by mouth) every evening at bed time. You will continue these injections 3 times a week and the daily oral medicine for up to 2 months if the therapy appears to be helping your disease.
  Interventions: Biological: sargramostim; Drug: thalidomide; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Biological: sargramostim — administered subcutaneously, generally well tolerated doses range from 50-500 ug/m2/day
  Other Names: GM-CSF
Drug: thalidomide — doses up to 400 mg/day
  Other Names: THALOMID
Procedure: conventional surgery — SOC care surgery
Procedure: neoadjuvant therapy — post radical prostatectomy

SUMMARY:
RATIONALE: Biological therapies, such as GM-CSF, may stimulate the immune system in different ways and stop tumor cells from growing. Thalidomide may stop the growth of prostate cancer by blocking blood flow to the tumor. Giving GM-CSF and thalidomide before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving GM-CSF together with thalidomide works in treating patients undergoing surgery for high-risk prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the impact of neoadjuvant sargramostim (GM-CSF) and thalidomide on pathologic response (histologic P0, margin positivity, capsular penetration), prostate-specific antigen (PSA) response, and other investigational endpoints in patients with high-risk prostate cancer undergoing prostatectomy.
* Determine the safety and feasibility of GM-CSF and thalidomide.

OUTLINE: This is an open-label study.

Patients receive sargramostim (GM-CSF) subcutaneously on days 1, 3, and 5 and oral thalidomide on days 1-5 or 1-7 in weeks 1-4. Treatment repeats every 4 weeks for 2 courses in the absence of unacceptable toxicity.

Patients undergo radical prostatectomy with bilateral pelvic lymphadenectomy at week 8 or 9.

PROJECTED ACCRUAL: A total of 29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate meeting any of the following criteria for high-risk disease:

  * Clinical stage II or III (T2b, T2c, or T3 with any grade or prostate-specific antigen [PSA])
  * Gleason score 7 (4+3 only) or ≥ 8 (any stage or PSA)
  * Serum PSA ≥ 10 ng/dL (any grade or stage)
  * Any stage, PSA, or Gleason score with ≥ 35% chance of biochemical failure at 5 years based on Kattan's nomogram
* No clinical evidence of CNS metastases
* No metastatic disease as demonstrated by radiological exam (CT scan, MRI, bone scan, x-ray) within 8 weeks of study entry
* Appropriate medical candidate for radical prostatectomy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Creatinine ≤ 2.0 mg/dL
* Granulocyte count ≥ 1,800/mm³
* Platelet count ≥ 100,000/mm³
* AST < 3 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL
* Fertile patients must use effective contraception during and for 4 weeks after completion of study treatment
* No active unresolved infection
* No pre-existing peripheral neuropathy > grade 1
* No known HIV positivity
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell carcinoma of the skin or controlled Ta transitional cell carcinoma of the bladder
* No known contraindication to sargramostim (GM-CSF) or thalidomide

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the prostate or pelvis
* No prior chemotherapy or hormonal therapy for prostate cancer
* No parenteral antibiotics within the past 7 days

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Garcia, MD, FACP, Principal Investigator — The Cleveland Clinic; Eric Klein, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GM-CSF Injections and Oral Thalidomide
Started | 28 (1 pt w/d consent. 1 pt found to have unresectable dx at time of sx and is exc. in tissue analysis.)
Completed | 26
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | GM-CSF Injections and Oral Thalidomide
Number analyzed (Participants) | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [44 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients P0 at Surgery
Description: Pathologic Complete Response is defined as complete eradication of tumor.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF Injections and Oral Thalidomide
Number analyzed (Participants) | 26
Participants | 0

2. Primary Outcome: Proportion of Patients With Negative Surgical Margins
Description: Presence or Absence of prostate cancer tissue at the sites of surgical resection. This is done by reviewing the entire specimen resected at the time or Radical Prostatectomy.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF Injections and Oral Thalidomide
Number analyzed (Participants) | 26
Participants | 0

3. Primary Outcome: Prostate-specific Antigen Response
Description: Number of subjects that achieved a PSA decline while on therapy. Any PSA decline while on treatment, compared with baseline PSA prior to study entry.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF Injections and Oral Thalidomide
Number analyzed (Participants) | 27
Participants | 22

4. Primary Outcome: Time to Clinical Progression
Description: Time to progression. WIth a median follow up of 32 months (12-51 months), 5 of 26 patients developed biochemical failure.
Time Frame: 32 months
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF Injections and Oral Thalidomide
Number analyzed (Participants) | 26
Participants | 5

ADVERSE EVENTS:
Arm/Group | GM-CSF Injections and Oral Thalidomide
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF Injections and Oral Thalidomide (N=27)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF Injections and Oral Thalidomide (N=27)
Constipation (Gastrointestinal disorders) | 17
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 15
Peripheral Neropathy (Nervous system disorders) | 7
Fatigue (General disorders) | 12
Solmnolene/Dizziness (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No